CLINICAL TRIAL: NCT04057651
Title: Study of Self-assessment Questionnaires Used in Hip and Knee Surgery
Brief Title: Hip and Knee Scores
Acronym: HIP-KNEE
Status: Completed | Type: Observational
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Other Study IDs: 2016_72; 2017-A01911-52 (Other: ID-RCB number, ANSM)
Record Dates: First submitted 2019-08-13; First posted 2019-08-15 (Actual); Last update posted 2020-09-16 (Actual); Status verified 2020-09

CONDITIONS: Hip Osteoarthritis; Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Hip; Osteoarthritis, Knee

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Hip osteoarthritis waiting for surgery
- Knee osteoarthritis waiting for surgery

SUMMARY:
Patient-reported outcome measures (PROMs) are currently used for evaluating orthopaedic procedures. Nevertheless, there is no consensus in the different studies, making them difficult to compare . The score mapping (or cross walk) is a statistical model for estimating a score associated with an unmeasured score.

Moreover , Minimal clinically important differences (MCID) is the smallest change in a treatment outcome that a patient would identify as important. The MCID is also not clearly identified for the French population for the hip and knee orthopaedic scores.

ELIGIBILITY:
Inclusion Criteria:

* Hip osteoarthritis (certified by standard radiographs)
* Knee osteoarthritis ( certified by standard radiographs)

Exclusion Criteria:

* BMI ≥ 40
* Systemic inflammatory disease
* Pregnant
* Surgery revision

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hip and knee patients waiting for hip and knee arthroplasty
Sampling Method: Non-Probability Sample
Enrollment: 800 (Actual)
Dates: Start 2018-08-28 (Actual); Primary Completion 2020-05-19 (Actual); Study Completion 2020-05-19 (Actual)

PRIMARY OUTCOMES:
Oxford Hip Score | The day Before surgery
  t is a 12-item patient-reported outcome measure designed to assess disability after surgery to the hip. Each item was scored between 0 and 4, with 4 been the best outcome per question producing overall scores running from 0 to 48(48 being the best outcome); > 41 is excellent, 34 - 41 is good,27 -33 as fair, and <27 is poor.
HOOS Score | The day Before surgery
  The HOOS (Hip disability and Osteoarthritis Outcome Score) is a patient questionnaire evaluating patients' feelings about their operated hip. It consists of 40 questions divided into 5 subgroups: pain, symptoms, daily living, quality of life, sports and recreational activities. Each category is scored on 100 points, 0 being the worse outcome and 100 the best outcome.
KOOS score | The day Before surgery
  Knee injury and Osteoarthritis Outcome Score (KOSS)
Oxford knee score | The day Before surgery
  Oxford Knee Score is a tool which measures 6 post operative items (pain,flexion contracture, extension lag, total range of flexion, alignment of varus and valgus,stability (antero-posterior and mediolateral). The scoring is: below 60 is poor, scoring 60-69 fair, scoring 70-79 good, 80-100 excellent.

SECONDARY OUTCOMES:
Oxford Hip Score | an average between 6 to 9 months after surgery
HOOS Score | an average between 6 to 9 months after surgery
KOOS score | an average between 6 to 9 months after surgery
Oxford knee Score | an average between 6 to 9 months after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Sophie Putman, MD, Principal Investigator — University Hospital, Lille
Locations (1):
- Hôpital Roger Salengro, CHU, Lille, France

REFERENCES:
- [Derived] Putman S, Preda C, Girard J, Duhamel A, Migaud H. Mapping and Crosswalk of the Oxford Hip Score and Different Versions of the Hip Disability and Osteoarthritis Outcome Score. Clin Orthop Relat Res. 2021 Jul 1;479(7):1534-1544. doi: 10.1097/CORR.0000000000001675. PMID 34128911
- [Derived] Putman S, Dartus J, Migaud H, Pasquier G, Girard J, Preda C, Duhamel A. Can the minimal clinically important difference be determined in a French-speaking population with primary hip replacement using one PROM item and the Anchor strategy? Orthop Traumatol Surg Res. 2021 May;107(3):102830. doi: 10.1016/j.otsr.2021.102830. Epub 2021 Jan 29. PMID 33524632